CLINICAL TRIAL: NCT07042178
Title: The Influence of Stress-inducing and Relaxing VR Content on Haematologic and Endocrinologic Blood Parameters in Healthy Participants - the 8baan Study
Brief Title: The Influence of Virtual Reality on Blood Parameters
Acronym: 8baan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Van Creveldkliniek (Other)
Responsible Party: Sponsor-Investigator, Van Creveldkliniek, Center for Benign Hematology, Thrombosis and Haemostasis, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 25U-0212; NL-009813 (Registry Identifier: onderzoekmetmensen.nl)
Record Dates: First submitted 2025-06-11; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Virtual Reality Pain Distraction; Endocrinology; Haematology
Keywords: Virtual reality; Stress-related biomarkers; Rollercoaster

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Arm A receives the Relax visit first and 3-5 weeks later the Rollercoaster Visit.
  Interventions: Other: Meditation video at the beach; Other: Rollercoaster video
- Arm B (Experimental): Arm B receives the Rollercoaster Visit first and 3-5 weeks later the Relax Visit.
  Interventions: Other: Meditation video at the beach; Other: Rollercoaster video

INTERVENTIONS:
Other: Meditation video at the beach — A virtual reality video consisting of a 5 minute meditation video at te beach.
Other: Rollercoaster video — A virtual reality video consisting of a five minute rollercoaster ride.

SUMMARY:
The goal of this study is to learn what the impact of exposure to virtual reality content is on the levels of stress-related blood values in healthy volunteers. The main question it aims to answer is:

* To compare the levels of stress-related biomarkers before and after relaxing VR-content (Relax Visit);
* To compare the levels of stress-related biomarkers before and after stress-inducing VR-content (Rollercoaster Visit).

Researchers will compare the Relax and Rollercoaster Visit to see if there is a relationship between the relaxing and stress-inducing VR content on stress-related blood values.

Participants will be asked to watch relaxing or stress-inducing VR content for approximately five minutes. Blood will be withdrawn before and after intervention. After 3-5 weeks the study visit will be repeated using the other VR content.

DETAILED DESCRIPTION:
Rationale: In recent years virtual reality (VR) has become increasingly popular in clinical setting, especially during blood sampling to enhance patient comfort and reduce anxiety. The immersion in a 360° fantasy world contributes to an effective way of distraction. During a medical procedure the patient is allowed to choose a VR interface that corresponds his liking. This can consist in relaxing content, like meditation video's or swimming with dolphins, or stress-inducing content, like a rollercoaster ride. The latter might be problematic due to its potential influence on stress levels. Many laboratory tests, like haematologic and endocrinologic markers can be influenced during an acute stress response. Normally, this physiological process ensures an effective energy metabolism when most needed. However, during a blood withdrawal using stress-inducing VR this is inconvenient as it could theoretically result in elevated or inaccurate laboratory tests. This might lead to additional blood draws, misdiagnoses and potential over- or undertreatment of patients. To the best of our knowledge, no previous research has assessed the accuracy of laboratory tests conducted on blood samples drawn during a VR rollercoaster experience.

Objective: To assess the impact of exposure to relaxing and stress-inducing virtual reality content on the levels of stress-related biomarkers in healthy individuals.

Study design: This is a monocentre pilot cross-over clinical trial. Study participants will be randomly assigned to one of the two arms. These arms determine the order of VR content exposure. The first arm will be exposed to relaxing VR content during the first study visit, during which blood will be drawn before and after the VR experience. Then, after an interval of 3-5 weeks, they will be exposed to stress-inducing VR content and blood will be drawn before and after. The second arm will do the study visits in the opposite order.

Study population: Healthy volunteers between the ages of 18 and 45 years with no medical history on haematologic, endocrinologic or cardiac disorders.

Intervention:

Participants will be exposed to stress-inducing and relaxing VR content during two separate study visits, the Relax Visit and the Rollercoaster Visit. Blood samples will be collected immediately before and after each VR session to measure changes in stress-related biomarkers. Additionally, objective stress levels measured by vital functions (e.g. heart rate, blood pressure) and subjective stress levels measured using a visual analogue scale (VAS) will be collected immediately pre- and post- VR exposure.

Main study parameters/endpoints:

The correlation between stress-related biomarkers (factor VIII activity, vWF ristocetin co-factor activity, copeptin (AVP), prolactin, thyroid stimulating hormone (TSH), cortisol and glucose) before and after relaxing and stress-inducing VR-content.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Participation includes two site visits, with an interval of 3 to 5 weeks. In both visits blood samples will be collected immediately before and after each VR session to measure changes in biomarkers. Additionally, objective stress levels measured by vital functions and subjective stress levels measured using a visual analogue scale will be collected immediately pre- and post- VR exposure. There are no benefits for participants. However, the results of this study may possibly benefit patients with haematological and endocrinological disorders regarding their comfort and anxiety during blood sampling and by reducing unnecessary extra sampling. Furthermore, it may benefit their treatment by optimizing the diagnostic process. Potential risks are the experience of motion-sickness during the VR experience and a blood withdrawal might be experienced as minimally painful for a very short amount of time. However, to minimalize this pain participants will apply a numbing cream one hour before the start of a study visit.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years old;
* Willing and able to provide written informed consent.

Exclusion Criteria:

* A history of motion- or cybersickness;
* Fear of needles;
* Any of the following haematological disorders:

  * Congenital or acquired haemophilia A;
  * Von Willebrand Disease.
* Any of the following endocrinological disorders:

  * Thyroid disorders (e.g. hypo/hyperthyroidism);
  * Cushing syndrome;
  * Adrenal insufficiency;
  * Diabetes mellitus type 1 or 2;
  * Central or nephrogenic AVP deficiency.
* A confirmed cardiac disorder;
* All types of epilepsy;
* Every form of medication, except for intermittent use of pain killers but not in the last week (e.g. paracetamol) and an intra-uterine device with or without contraceptive;
* Pregnancy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The effect of relaxing VR content on von Willebrand ristocetin co-factor activity | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to relaxing VR content (approximately 10 minutes later)
  The difference between von Willebrand ristocetin co-factor activity before and after relaxing VR content (beach meditation video) is measured.
The effect of stress-inducing VR content on von Willebrand ristocetin co-factor activity | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to stress-inducing VR content (approximately 10 minutes later)
  The difference between von Willebrand ristocetin co-factor activity before and after stress-inducing VR content (rollercoaster ride) is measured.
The correlation between relaxing and stress-inducing VR content on von Willebrand ristocetin co-factor activity | From baseline to the end of the second VR video (type is depending on assigned arm) (approximately 3-5 weeks later)
  The relationship between relaxing (beach meditation video) and stress-inducing VR content (rollercoaster video) for von Willebrand ristocetin co-factor activity is assessed.
The effect of relaxing VR content on FVIII activity | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to relaxing VR content (approximately 10 minutes later)
  The difference between FVIII activity before and after relaxing VR content (beach meditation video) is measured.
The effect of stress-inducing VR content on FVIII activity | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to stress-inducing VR content (approximately 10 minutes later)
  The difference between FVIII activity before and after stress-inducing VR content (rollercoaster ride) is measured.
The correlation between relaxing and stress-inducing VR content on FVIII activity | From baseline to the end of the second VR video (type is depending on assigned arm) (approximately 3-5 weeks later)
  The relationship between relaxing (beach meditation video) and stress-inducing VR content (rollercoaster video) for FVIII activity is assessed.
The effect of relaxing VR content on copeptin | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to relaxing VR content (approximately 10 minutes later)
  The difference between copeptin before and after relaxing VR content (beach meditation video) is measured.
The effect of stress-inducing VR content on copeptin | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to stress-inducing VR content (approximately 10 minutes later)
  The difference between copeptin before and after stress-inducing VR content (rollercoaster ride) is measured.
The correlation between relaxing and stress-inducing VR content on copeptin | From baseline to the end of the second VR video (type is depending on assigned arm) (approximately 3-5 weeks later)
  The relationship between relaxing (beach meditation video) and stress-inducing VR content (rollercoaster video) for copeptin is assessed.
The effect of relaxing VR content on prolactin | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to relaxing VR content (approximately 10 minutes later)
  The difference between prolactin before and after relaxing VR content (beach meditation video) is measured.
The effect of stress-inducing VR content on prolactin | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to stress-inducing VR content (approximately 10 minutes later)
  The difference between prolactin before and after stress-inducing VR content (rollercoaster ride) is measured.
The correlation between relaxing and stress-inducing VR content on prolactin | From baseline to the end of the second VR video (type is depending on assigned arm) (approximately 3-5 weeks later)
  The relationship between relaxing (beach meditation video) and stress-inducing VR content (rollercoaster video) for prolactin is assessed.
The effect of relaxing VR content on thyroid stimulating hormone (TSH) | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to relaxing VR content (approximately 10 minutes later)
  The difference between TSH before and after relaxing VR content (beach meditation video) is measured.
The effect of stress-inducing VR content on TSH | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to stress-inducing VR content (approximately 10 minutes later)
  The difference between TSH before and after stress-inducing VR content (rollercoaster ride) is measured.
The correlation between relaxing and stress-inducing VR content on TSH | From baseline to the end of the second VR video (type is depending on assigned arm) (approximately 3-5 weeks later)
  The relationship between relaxing (beach meditation video) and stress-inducing VR content (rollercoaster video) for TSH is assessed.
The effect of relaxing VR content on cortisol | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to relaxing VR content (approximately 10 minutes later)
  The difference between cortisol before and after relaxing VR content (beach meditation video) is measured.
The effect of stress-inducing VR content on cortisol | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to stress-inducing VR content (approximately 10 minutes later)
  The difference between cortisol before and after stress-inducing VR content (rollercoaster ride) is measured.
The correlation between relaxing and stress-inducing VR content on cortisol | From baseline to the end of the second VR video (type is depending on assigned arm) (approximately 3-5 weeks later)
  The relationship between relaxing (beach meditation video) and stress-inducing VR content (rollercoaster video) for cortisol is assessed.
The effect of relaxing VR content on glucose | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to relaxing VR content (approximately 10 minutes later)
  The difference between glucose before and after relaxing VR content (beach meditation video) is measured.
The effect of stress-inducing VR content on glucose | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to stress-inducing VR content (approximately 10 minutes later)
  The difference between glucose before and after stress-inducing VR content (rollercoaster ride) is measured.
The correlation between relaxing and stress-inducing VR content on glucose | From baseline to the end of the second VR video (type is depending on assigned arm) (approximately 3-5 weeks later)
  The relationship between relaxing (beach meditation video) and stress-inducing VR content (rollercoaster video) for glucose is assessed.

SECONDARY OUTCOMES:
The effect of relaxing VR-content on blood pressure | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to relaxing VR content (approximately 10 minutes later)
  The difference before and after relaxing VR-content (beach meditation video) on blood pressure
The effect of stress-inducing VR-content on blood pressure | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to stress-inducing VR content (approximately 10 minutes later)
  The difference before and after stress-inducing VR-content (rollercoaster ride video) on blood pressure
The correlation between relaxing and stress-inducing VR content on blood pressure | From baseline to the end of the second VR video (type is depending on assigned arm) (approximately 3-5 weeks later)
  The relationship between relaxing (beach meditation video) and stress-inducing VR content (rollercoaster video) for blood pressure is assessed.
The effect of relaxing VR-content on temperature | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to relaxing VR content (approximately 10 minutes later)
  The difference before and after relaxing VR-content (beach meditation video) on temperature
The effect of stress-inducing VR-content on temperature | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to stress-inducing VR content (approximately 10 minutes later)
  The difference before and after stress-inducing VR-content (rollercoaster ride video) on temperature
The correlation between relaxing and stress-inducing VR content on temperature | From baseline to the end of the second VR video (type is depending on assigned arm) (approximately 3-5 weeks later)
  The relationship between relaxing (beach meditation video) and stress-inducing VR content (rollercoaster video) for temperature is assessed.
The effect of relaxing VR-content on heart rate | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to relaxing VR content (approximately 10 minutes later)
  The difference before and after relaxing VR-content (beach meditation video) on heart rate
The effect of stress-inducing VR-content on heart rate | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to stress-inducing VR content (approximately 10 minutes later)
  The difference before and after stress-inducing VR-content (rollercoaster ride video) on heart rate
The correlation between relaxing and stress-inducing VR content on heart rate | From baseline to the end of the second VR video (type is depending on assigned arm) (approximately 3-5 weeks later)
  The relationship between relaxing (beach meditation video) and stress-inducing VR content (rollercoaster video) for heart rate is assessed.
The effect of relaxing VR-content on respiratory rate | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to relaxing VR content (approximately 10 minutes later)
  The difference before and after relaxing VR-content (beach meditation video) on respiratory rate
The effect of stress-inducing VR-content on respiratory rate | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to stress-inducing VR content (approximately 10 minutes later)
  The difference before and after stress-inducing VR-content (rollercoaster ride video) on respiratory rate
The correlation between relaxing and stress-inducing VR content on respiratory rate | From baseline to the end of the second VR video (type is depending on assigned arm) (approximately 3-5 weeks later)
  The relationship between relaxing (beach meditation video) and stress-inducing VR content (rollercoaster video) for respiratory rate is assessed.
The effect of relaxing VR content on subjective stress reported by participant | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to relaxing VR content (approximately 10 minutes later)
  Subjective stress, measured by a visual analogue scale (VAS) (scale 0-10 made visual using different faces; 0 being no stress, 10 being the worst stress a person can imagine), during relaxing VR content (beach meditation video).
The effect of stress-inducing VR content on subjective stress reported by participant | From baseline (5 minutes before start of the VR content during a study visit) to the end of the exposure to stress-inducing VR content (approximately 10 minutes later)
  Subjective stress, measured by a visual analogue scale (VAS) (scale 0-10 made visual using different faces; 0 being no stress, 10 being the worst stress a person can imagine), during relaxing VR content (rollercoaster ride video).

CONTACTS AND LOCATIONS:
Overall Officials: Corien L. Eckhardt, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Centre Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
After finishing the project, the data package will be stored at the UMC Utrecht Research Folder Structure and is under the responsibility of the Principal Investigator of the research group. The metadata will be available in the UMCU repository (DataverseNL).
  As the data is privacy-sensitive, we publish the descriptive metadata in the data repository with a description of how a data request can be made (by sending an email to the corresponding author). In the event that peers like to reuse our data this can only be granted if the research question is in line with the original informed consent signed by the study participants. Every application therefore will be screened upon this requirement. If granted, a data usage agreement is signed by the receiving party.
Supporting Information: CSR